CLINICAL TRIAL: NCT02847377
Title: Exploratory Phase 0/1 of Positron Emission Tomography (PET) Imaging Agent [18F]-ODS2004436 as a Marker of EGFR Mutation in Subjects With NSCLC
Brief Title: A Positron Emission Tomography (PET) Imaging Agent [18F]-ODS2004436 as a Marker of EGFR Mutation in Subjects With NSCLC
Acronym: IMKRUN 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IMK RUN 2
Record Dates: First submitted 2016-07-12; First posted 2016-07-28 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2019-11

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [18F]-ODS2004436 (Experimental): Two TEP will be performed with the radiotracer [18F]-ODS2004436
  Interventions: Other: Injection of [18F]-ODS2004436 radiotracer

INTERVENTIONS:
Other: Injection of [18F]-ODS2004436 radiotracer

SUMMARY:
The development of biomarkers will lead the dynamic of personalized medicine and fill the unsatisfied needs in oncology for prediction of therapeutic response.

Molecular imaging enables non invasive quantification of biomarkers. The development of molecular imaging biomarkers is closely related to the development of therapeutic molecules. Among the potential targets, kinases offer a lot of advantages: (i) they play a central role in cellular regulation, (ii) numerous kinase-specific small molecule libraries exist in biotech and pharma industry, (iii) several kinase-targeted therapies are used in clinic (imatinib, sorafenib, sunitinib…) with application across a variety of therapeutic indications. Among the imaging technologies, the Positron Emission Tomography (PET) is the most sensitive and dedicated to evaluate small molecules. However few radiotracers are available and their specificity limits their clinical use. The IMAkinib® approach is an innovative method proposed to develop new PET radiotracers adapted to current medical and economical challenges.

The epidermal growth factor receptor (EGFR) is an established target for the treatment of advanced non-small cell lung cancer (NSCLC). The EGFR tyrosine kinase inhibitors (TKIs) Gefitinib (Iressa®), erlotinib (Tarceva®) and afatinib (Giotrif®) have already been approved for treatment of NSCLC harboring EGFR activating mutations (L858R or del exon 19). Unfortunately the majority of patients will develop a resistance to the TKI in the long term (6-12 months). If the mechanism of resistance is not yet fully characterized, most patients (50%) will acquire an additional T790M mutation of EGFR. TKI PET-imaging can provide a tool to determine and predict responsiveness to EGFR TKI in vivo. That is why, the investigators have selected and radiolabeled (18-Fluor) a compound targeting specifically EGFR mutated ([18F]-ODS2004436) which was further evaluated in a preclinical imaging study to determine the feasibility of TKI-PET. The investigators proved in vivo that [18F]-ODS2004436 a compound is a good candidate to evaluate the EGFR activity in human lung tumours using PET imaging.

ELIGIBILITY:
Inclusion Criteria:

* more than 18 years,
* Willing and able to sign written informed consent,
* Histologically confirmed diagnosis of adenocarcinoma NSCLC:

  1. positive mutated KRas homogeneous population for EGFR Wild type (WT) patients (exclusive with EGFR mutation)
  2. EGFR activating mutation (All mutations: 719, 790, 861, 858 or del exon 19 and exon 20),
* Patient with EGFR mutation will be sensitive to TKI
* Treatment naïve patients,
* Performance status ≤ 2 on the Eastern Cooperative Oncology Group (ECOG) criteria,
* No concomitant prescriptions including cyclosporin A, valproic acid, phenobarbital, phenytoin, ketoconazole,
* Adequate hematologic (ANC count ≥ 1,500/uL, platelet count ≥ 100,000/mm3), hepatic (bilirubin level ≤ 1.5 mg/dL, Transaminase (AST/ALT) ≤ 80 IU/L), and renal (creatinine concentration ≤ 1.5 mg/dL) function,
* Patients with brain metastasis are allowed unless there were clinically significant neurological symptoms or signs.

Exclusion Criteria:

* Known severe hypersensitivity to Gefitinib or Afatinib or any of the tablet excipients,
* Inability to swallow tablets,
* Other coexisting malignant disease,
* Concomitant use of phenytoin, carbamazepine, rifampicin, barbiturates, or St John's wort; severe or uncontrolled systemic disease; clinically active interstitial lung disease (except uncomplicated lymphangitic carcinomatosis),
* Female subjects who are pregnant, breast-feeding or male or female patients of reproductive potential who are not employing an effective method of birth control,
* Subjects under guardianship, curators or judicial protection

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-09-27 (Actual); Primary Completion 2016-09-27 (Actual); Study Completion 2019-03-19 (Actual)

PRIMARY OUTCOMES:
Evaluation of sensibility of [18F] ODS2004436 | 1 day
  Sensibility will be evaluated by positron emission tomography (PET) performed on EGFR mutant patient
Evaluation of specificity of [18F] ODS2004436 | 1 day
  Specificity will be evaluated by positron emission tomography (PET) performed on EGFR wild type patient

OTHER OUTCOMES:
Security | 10 days
  A follow up visit will be performed 3 days after each PET has been performed in order to register adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Pierre FUMOLEAU, Pr, Study Director — Centre Georges Francois Leclerc
Locations (1):
- CGFL, Dijon, France